CLINICAL TRIAL: NCT03996746
Title: Prospective Evaluation of Serum Klotho, a Novel Biomarker, as a Predictor of Progression of Cardiovascular Calcification (CVC) in Chronic Kidney Disease (CKD)
Brief Title: Evaluation of Serum Klotho as a Predictor of Progression of Cardiovascular Calcification in Chronic Kidney Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: XH-19-003
Record Dates: First submitted 2019-06-23; First posted 2019-06-25 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Chronic Kidney Disease
Keywords: Klotho; Cardiovascular Calcification
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-dialysis Group: non-dialysis patients with CKD 2-5
  Interventions: Diagnostic Test: No intervention
- Hemodialysis Group: patients with CKD 5 under hemodialysis for more than 3 months
  Interventions: Diagnostic Test: No intervention

INTERVENTIONS:
Diagnostic Test: No intervention — No intervention

SUMMARY:
This prospective observational study aims to investigate the relationship between CVC and serum Klotho for renal function correction in patients with different CKD stages

DETAILED DESCRIPTION:
In this study, we plan to enroll 400 non-dialysis patients with CKD 2-5 and 300 maintenance hemodialysis patients. Participants will receive coronary artery computed tomography (CT) scanning to detect the extent and the severity of CVC. Follow-up is scheduled at 0, 6, 12, 18, and 24 months and will consist the following: routine physical examinations, standard lab panels (blood routine, liver/kidney functions, tests of the coagulation system, etc.), total calcium, phosphate, parathyroid hormone (PTH), serum 25(OH) vitamin D, fibroblast growth factor-23 (FGF-23) and coronary artery computed tomography (CT).

The purpose of this study was to clarify the relationship between CVC in patients with different CKD stages and serum Klotho for renal function correction, and to clarify that Klotho can be used as an early biomarker for CVC in patients with CKD, so as to predict the occurrence and progress of CVC.

ELIGIBILITY:
Inclusion Criteria:

1. age over 18 years old, regardless of gender
2. non-dialysis patients with CKD 2-5, or patients with CKD 5 under hemodialysis for more than 3 months

Exclusion Criteria:

1. life expectancy < 2 years
2. severe complications of heart, lung, liver or brain
3. primary hyperparathyroidism
4. malignant tumor
5. pregnant or breastfeeding
6. contraindications to CT examination
7. unwilling or unable to comply with the research protocol

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Two different populations will be selected. First group will be non-dialysis patients with CKD 2-5. Second group will be patients with CKD 5 under hemodialysis for more than 3 months.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2019-06-25 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
The relationship between CVC and serum Klotho | From date of enrollment until the end of study, assessed up to 24 months
  To clarify the relationship between CVC and serum Klotho for renal function correction in patients with different CKD stages, and to clarify that Klotho can be used as an early biomarker for CVC in patients with CKD, so as to predict the occurrence and progress of CVC

SECONDARY OUTCOMES:
The sensitivity and specificity of serum Klotho in the detection of CVC | From date of enrollment until the end of study, assessed up to 24 months
  To evaluate the sensitivity and specificity of serum Klotho in the detection of cardiovascular calcification and to clarify its status as a biomarker of calcification

CONTACTS AND LOCATIONS:
Overall Officials: Wei LU, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Xinhua Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No